CLINICAL TRIAL: NCT06556043
Title: Investigating the Effects of Transcranial Direct Current Stimulation (tDCS) to Different Brain Regions on Ankle Tracking Motor Learning, Motor Adaptation, and Brain Connectivity in Healthy Middle-aged and Older Adults and Patients With Subcortical Stroke
Brief Title: Investigating the Effects of Transcranial Direct Current Stimulation to Different Brain Regions on Ankle Tracking Motor Learning, Motor Adaptation, and Brain Connectivity in Healthy Middle-aged and Older Adults and Patients With Subcortical Stroke
Acronym: tDCS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 202212150DINB
Record Dates: First submitted 2023-02-21; First posted 2024-08-15 (Actual); Last update posted 2024-08-19 (Actual); Status verified 2024-02

CONDITIONS: Transcranial Direct Current Stimulation; Ankle; Motor Learning; Adaptation; Brain Structure; Brain Connectivity; Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- cM1 stimulation group (Experimental): cM1= primary motor cortex (M1) contralateral to the moving leg
  Interventions: Other: cM1 transcranial direct current stimulation
- cPPC stimulation group (Experimental): cPPC= posterior parietal cortex (PPC) contralateral to the moving leg
  Interventions: Other: cPPC transcranial direct current stimulation
- iCBM stimulation group (Experimental): iCBM= cerebellar cortex ipsilateral to the moving leg
  Interventions: Other: iCBM transcranial direct current stimulation
- Sham group (Sham Comparator)
  Interventions: Other: sham transcranial direct current stimulation

INTERVENTIONS:
Other: cM1 transcranial direct current stimulation — During the 5-day skill acquisition phase, all participants will undertake a 20-minute session of learning a sequential ankle tracking task with their non-dominant (for healthy adults) or affected (for patients with stroke) foot each day, using a custom-built ankle tracking system. The cM1 group will receive AtDCS stimulation at 2 mA during acquisition phase.
  Arms: cM1 stimulation group
Other: cPPC transcranial direct current stimulation — During the 5-day skill acquisition phase, all participants will undertake a 20-minute session of learning a sequential ankle tracking task with their non-dominant (for healthy adults) or affected (for patients with stroke) foot each day, using a custom-built ankle tracking system. The cPPC group will receive AtDCS stimulation at 2 mA during acquisition phase.
  Arms: cPPC stimulation group
Other: iCBM transcranial direct current stimulation — During the 5-day skill acquisition phase, all participants will undertake a 20-minute session of learning a sequential ankle tracking task with their non-dominant (for healthy adults) or affected (for patients with stroke) foot each day, using a custom-built ankle tracking system. The iCBM group will receive AtDCS stimulation at 2 mA during acquisition phase.
  Arms: iCBM stimulation group
Other: sham transcranial direct current stimulation — For the Sham group, the montages of the paired electrode placements will be randomly selected from the other three pairs using blocks of size 3, so that the three types of montages will have equal opportunities to be used in the Sham group. The intensity will be set at 0 mA for the Sham group. There will be a 30-second ramp-up for the Sham group. Once the current reaches 2 mA in the ramp-up period, it will drop to 0 mA for the entire 20 minutes during learning for the Sham group.
  Arms: Sham group

SUMMARY:
Ankle control is essential to safe over-ground navigation for humans. Middle- aged and older adults and patients with stroke whose ankle control is poor often lose their balance or fall. Transcranial direct current stimulation (tDCS) is an emerging non-invasive brain stimulation technology that has great potential to be applied to neurorehabilitation; however, the optimization of its applications still needs further studies. The aims of this project are to compare the effects of anodal tDCS (AtDCS) applied to the primary motor cortex (M1) contralateral to the moving leg (cM1), posterior parietal cortex (PPC) contralateral to the moving leg (cPPC), and cerebellar cortex (CBM) ipsilateral to the moving leg (iCBM) on motor learning, motor adaptation, and brain connectivity in healthy middle-aged and older adults and hemiparetic patients with chronic subcortical stroke.

ELIGIBILITY:
Inclusion Criteria: Part 1: healthy middle-aged and older adults

1. age between 40 and 80 years old
2. intact cognitive function (MMSE ≧ 27)
3. normal ankle dorsiflexor and plantarflexor strength (manual muscle strength testing= 5) and passive range of motion (ankle dorsiflexion ≧10 degrees; ankle plantarflexion ≧ 45 degrees)
4. corrected far vision ≥ 0.8 (Landolt C test) and uncorrected near vision ≥ 0.04 (Comprehensive Color Blindness Checklist)

Exclusion Criteria: Part 1: healthy middle-aged and older adults

1. having any contraindications for MRI or tDCS;
2. serious or uncontrolled systematic diseases;
3. symptoms or history of neurological diseases, including transient ischemic attack, stroke, epilepsy, history of abnormal electroencephalogram (EEG), meningitis, encephalitis, brain tumors, brain surgery, and sensory disorders, etc.;
4. severe musculoskeletal problems that would affect lower limb functions;
5. visual spatial perception disorders and hearing loss;
6. color blindness;
7. depression and psychiatric disorders;
8. use of any medication that could affect the central nervous system function;
9. drug, substance, or alcohol addiction;
10. those participating in research involving invasive or non-invasive brain stimulation;
11. those deemed unsuitable for MRI or tDCS after evaluation by the attending physician;
12. those affiliated with any research-conducting institution.

Inclusion Criteria: Part 2: patients with chronic subcortical stroke

1. aged between 40 and 80 years old;
2. intact cognitive function (MMSE ≥ 27);
3. first-ever onset of subcortical stroke occurring at least 3 months prior to enrollment, with brain lesions involving unilateral subcortical regions only;
4. hemiplegic or hemiparetic;
5. no spatial neglect;
6. able to actively perform at least 5 degrees of ankle dorsiflexion and 10 degrees of ankle plantarflexion with the affected ankle;
7. no excessive spasticity;
8. no severe contracture (passive range of motion ≥ 10 degrees for ankle dorsiflexion and ≥ 20 degrees for ankle plantarflexion) in the affected leg;
9. mild-to moderate disability;
10. can walk independently or under supervision without assistance;
11. corrected far vision ≥ 0.8 (Landolt C test) and uncorrected near vision ≥ 0.04 (Comprehensive Color Blindness Checklist.)

Exclusion Criteria: Part 2: patients with chronic subcortical stroke The exclusion criteria will be the same as those listed for healthy participants described in Part 1 except for items (3) and (4). Item (3) will be changed to "(3a) symptoms or history of other neurological diseases, including epilepsy, history of abnormal EEG, meningitis, encephalitis, brain tumors, brain surgery, and sensory disorders, etc." and item (4) will be changed to "(4a) severe musculoskeletal problems of the non-hemiparetic limbs that would affect mobility functions".

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-07-09 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Change of mean RMSE value of ankle tracking performances | 1 week
  Using a custom-built ankle tracking system
Change of Brain MRI data acquisition | 1 week
  Structural images: T1- and T2 weighted imaging, fluid attenuation inversion recovery (FLAIR) images, and diffusion spectrum image (DSI) Functional image: Resting-state functional MRI (rs-fMRI) images using a T2* gradient echo, echo-planar sequence.

SECONDARY OUTCOMES:
Fall histories | 1 week
  Fall Efficacy Scale (16~64 points, the higher score, the worsen outcome)
Attention | 1 week
  language-free Color Trail Test- Part 1
Muscle strength of bilateral ankle dorsiflexors and plantarflexors | 1 week
  Measured with a hand-held dynamometer
Mobility | 1 week
  "Timed "Up and Go" test, four square step test
Single-task gait | 1 week
  Measured with the GAITRite
Sensory and motor functions of patients with stroke | 1 week
  Fugl-Meyer Assessment
Balance | 1 week
  One-leg stance

CONTACTS AND LOCATIONS:
Overall Officials: Pei-Fang Tang, PhD, Principal Investigator — School and Graduate Institute of Physical Therapy, College of Medicine, National Taiwan University, Taiwan
Locations (1):
- School and Graduate Institute of Physical Therapy, National Taiwan University, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No